CLINICAL TRIAL: NCT03819400
Title: Evaluation of Kidney Graft's Fibrosis With Real Time Shear-wave Elastography
Acronym: Elastogreffe
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI18-Elastogreffe
Record Dates: First submitted 2019-01-25; First posted 2019-01-28 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Kidney Graft
Keywords: kidney graft; fibrosis; elastography
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Kidney graft's fibrosis is correlated with prognostic of kidney's graft, wathever the initial etiology. Actually, that evaluation is based on histologic score of Banff FI/AT (0 to III). It is obtained thanks to punction-biopsy, which is invasive and can lead complications. This exam is systematic on M3 of the transplantation.

Tissue's fibrosis is a proliferation of extracellular matrix, leading to an increase of fibrosed tissue rigidity.

Elastography is an ultrasound technique allowing evaluation of tissues' rigidity.

The purpose is the validation of elastograhpy, innovative and non -invasive technique, and more specifically Shear Wave Elastography (SWE). For this, strain ratio (SR) could improve intra-operator variability and estimate fibrosis' degree of kidney's graft.

DETAILED DESCRIPTION:
Kidney graft's fibrosis is correlated with prognostic of kidney's graft, wathever the initial etiology. Actually, that evaluation is based on histologic score of Banff FI/AT (0 to III). It is obtained thanks to punction-biopsy, which is invasive and can lead complications. This exam is systematic on M3 of the transplantation.

Tissue's fibrosis is a proliferation of extracellular matrix, leading to an increase of fibrosed tissue rigidity.

Elastography is an ultrasound technique allowing evaluation of tissues' rigidity.

The purpose is the validation of elastograhpy, innovative and non -invasive technique, and more specifically Shear Wave Elastography (SWE). For this, strain ratio (SR) could improve intra-operator variability and estimate fibrosis' degree of kidney's graft.

ELIGIBILITY:
Inclusion Criteria:

* Kidney-transplanted patient, whatever kind of organ donation ( alive donor, deceased donor included extended criteria Maastricht 2 or 3)
* More than 18 years-old

Exclusion Criteria:

* Dual kidney graft
* Hydronephrosis / urinary obstacle
* Pathologies with an intrinsic compression on the graft
* Stenosis hemodynamically significant of graft artery (lengthening of Systolic Ascent Time > 70 ms)
* Contra-indication to systematical punction-biopsy on Month 3 :

  * Ischemia of post-transplanted graft
  * Alive donor HLA identical
  * Hemostasis disorder or unable to stop antiaggregant or anticoagulant
  * Hydronephrosis / urinary obstacle
* Opposition to use the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney-transplanted patient
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
measure of shear wave elastography | 3 months
  Evaluation of shear wave elastography real time as biomarker of kidney graft's fibrosis

SECONDARY OUTCOMES:
Strain Ratio measure | 3 months
  - Intra-operator variability of Strain Ratio measure

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Tours, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided